CLINICAL TRIAL: NCT02066194
Title: Electroacupuncture Analgesia for Endoscopic Ultrasound (EUS): a Prospective, Randomized, Double-blinded, Sham-controlled Study
Brief Title: Electroacupuncture Analgesia for EUS: a Randomized Controlled Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Anthony Teoh, MD, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRE-2011.324
Record Dates: First submitted 2014-02-16; First posted 2014-02-19 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Patients Undergoing Endoscopic Ultrasound
MeSH Terms: interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Electroacupuncture (Active Comparator): Patients randomized to the experimental group will receive EA at acupoints relevant to the treatment of abdominal pain and anxiety. Selection of these acupoints is based on a consensus between the acupuncturist of the study (Leung WW) and several professors of the Diploma Course of Clinical Acupuncture of the School of Professional and Continuing Education, University of Hong Kong.
  Interventions: Procedure: Electroacupuncture
- Sham Acupuncture (Placebo Comparator): Patients randomized to the control group will receive Sham acupuncture with sterile blunt-tip needles
  Interventions: Procedure: Electroacupuncture

INTERVENTIONS:
Procedure: Electroacupuncture

SUMMARY:
Endoscopic ultrasound (EUS) has evolved to become an important diagnostic tool and its interventional role is rapidly expanding. In order to improve patient's comfort and satisfaction during and after procedure, the use of sedation is usually recommended. However, sedation may be associated with serious adverse events of including hypotension, aspiration and respiratory depression. Moreover, the cost of performing the procedure would be increased due to the costs of the medications and the need of additional personnel in monitoring of the patient. As a result, the drive to seek alternative and safer approaches of pain-relief during EUS is ever present. Electroacupuncture (EA) has been used in Traditional Chinese Medicine (TCM) for more than 2000 years. The benefits and success of EA in treatment of acute and chronic pain of various origins have been well-recognised. Many researches have been performed to address the role of EA in treating pain and anxiety during OGD and colonoscopy. However, only limited data is availabe in the Chinese and the Western literature concerning the use of EA in EUS. Therefore it is worthwhile to conduct a well-designed study to evaluate the role of EA in treating pain during EUS.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients (aged between 18 and 80 years) undergoing first-time elective day-case EUS, patients with American Society of Anesthesiologists (ASA) grading I-II, and informed consent available.

Exclusion Criteria:

* Patients with previous experience of acupuncture, patients with coagulopathy, patients with previous history of upper gastrointestinal surgery, patients who are diagnosed with irritable bowel syndrome according to Rome III criteria, 12 patients with chronic pain syndrome, patients with psychiatric disorder, patients with poor cognitive function, patients with renal impairment, patients with obstructive sleep apnea syndrome, patients with cardiac arrhythmias, patients with cardiac pacemaker, patients who are pregnant, and patients who are allergic to the acupuncture needles or Propofol/Alfentanil.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2014-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Consumption of propofol | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Teoh AYB, Chong CCN, Leung WW, Chan SKC, Tse YK, Ng EKW, Lai PBS, Wu JCY, Lau JYW. Electroacupuncture-reduced sedative and analgesic requirements for diagnostic EUS: a prospective, randomized, double-blinded, sham-controlled study. Gastrointest Endosc. 2018 Feb;87(2):476-485. doi: 10.1016/j.gie.2017.07.029. Epub 2017 Jul 24. PMID 28750840